CLINICAL TRIAL: NCT03024567
Title: Effects of Increased Salt Intake on Energy Metabolism in Healthy Volunteers - a Randomized Clinical Study
Brief Title: Randomized Study on Salt Intake and Energy Metabolism
Acronym: TS4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Anja Maehler, Principle Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Tissue Salt 4
Record Dates: First submitted 2017-01-13; First posted 2017-01-19 (Estimated); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Healthy
Keywords: Calorimetry; Blood pressure; Immunophenotyping; Gut microbial composition
MeSH Terms: interventions — Salts

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salt (Active Comparator): 6 grams sodium chloride per day for 14 days
  Interventions: Dietary Supplement: Salt
- Placebo (Placebo Comparator): 6 grams gelatine per day for 14 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Salt — 10 capsules daily for 14 days
  Arms: Salt
Dietary Supplement: Placebo — 10 capsules daily for 14 days
  Arms: Placebo

SUMMARY:
To perform a randomized, double-blind clinical study on the effects of an increased salt intake on metabolic, cardiovascular and immunological parameters and the gut microbiota

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18 - 50 years
* Body mass index 18.5 - 29.9 kg/m2

Exclusion Criteria:

* Clinically relevant heart, lung, liver, and kidney diseases
* Current or chronic infection
* Habitual use of probiotics or dietary supplements
* Pregnancy, lactation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Dietary induced thermogenis (%) | 14 days
  Decrease of dietary induced thermogenis after salt vs. placebo

SECONDARY OUTCOMES:
Systolic blood pressure (mmHg) | 14 days
  Increase of systolic blood pressure after salt vs. placebo
Lymphocytic pro-inflammatory mediators | 14 days
  Increase of lymphocytic pro-inflammatory mediators after salt vs. placebo
Gut microbiome | 14 days
  Change of gut microbiome composition after salt vs. placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Experimental and Clinical Research Center, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mahler A, Klamer S, Maifeld A, Bartolomaeus H, Marko L, Chen CY, Forslund SK, Boschmann M, Muller DN, Wilck N. Increased Salt Intake Decreases Diet-Induced Thermogenesis in Healthy Volunteers: A Randomized Placebo-Controlled Study. Nutrients. 2022 Jan 7;14(2):253. doi: 10.3390/nu14020253. PMID 35057434